CLINICAL TRIAL: NCT03222258
Title: Change of Quality of Life, Treatment Decision and Utilization of Health Care Depending on the Use of Palliative Care in Adult and Pediatric Patients With Advanced Stage of Cancer: a Prospective Cohort Study
Brief Title: Prospective Cohort Study Depending on the Use of Palliative Care for Advanced Stage of Cancer Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); National Cancer Center, Korea (Other Government); Kyunghee University Medical Center (Other); Severance Hospital (Other); Gyeongsang National University Hospital (Other); Chungnam National University Hospital (Other); Chonbuk National University Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Daegu Fatima Hospital (Other); Chonnam National University Hospital (Other); Keimyung University Dongsan Medical Center (Other); Hallym University Medical Center (Other); Asan Medical Center (Other); National Evidence-Based Healthcare Collaborating Agency (Other Government); National Institute of Health, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Young Ho Yun, Clinical Professor, Seoul National University Hospital
Other Study IDs: HC15C1391-2
Record Dates: First submitted 2017-06-05; First posted 2017-07-19 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Stage IV Breast Cancer; Stage IV Pancreatic Cancer; Stage IV Colon Cancer; Stage IV Gastric Cancer; Stage IV Lung Cancer; Stage IV Liver Cancer; Malignant Hematologic Neoplasm; Biliary Cancer Metastatic; Pediatric Leukemia; Pediatric Lymphoma; Pediatric Brain Tumor; Pediatric Solid Tumor
Keywords: Palliative Care; Quality of Life; Prospective Cohort Study; Treatment decision; Utilization of health care
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Stomach Neoplasms; Lung Neoplasms; Liver Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Early palliative care for adult: Being referred to palliative care team before totally terminating their chemotherapy among adult participants.
  Interventions: Behavioral: Early palliative care; Behavioral: Routine hospice care
- Routine hospice care for adult: Being referred to palliative care team when their last chemotherapy is ended among adult participants.
  Interventions: Behavioral: Routine hospice care
- Unused palliative care for adult: haven't been under the palliative care among adult participants
- Palliative care for pediatrics: receiving the palliative care among pediatric participants
  Interventions: Behavioral: Early palliative care; Behavioral: Routine hospice care
- Unused palliative care for pediatrics: haven't received the palliative care among pediatric participants

INTERVENTIONS:
Behavioral: Early palliative care — Palliative Care Team provide a self-learning booklet, medical treatment and consultation about Advance Care Planning with chemotherapy by oncologist.
  Groups: Early palliative care for adult; Palliative care for pediatrics
Behavioral: Routine hospice care — Palliative Care Team provide a routine hospice care the same as other patients who doesn't participate this study after the chemotherapy is totally terminated
  Groups: Early palliative care for adult; Palliative care for pediatrics; Routine hospice care for adult

SUMMARY:
This study evaluates the change of quality of life, treatment decision and utilization of health care depending on the use of palliative care in advanced cancer patients by a prospective cohort study. Participants will be separated into different groups by their intentions for using palliative care. Every participant will carry out the questionnaire per 3 months. This cohort study will be ended a year after each participant enrolls. However, if the participant didn't survive during this study, the caregivers will be asked to fill out additional questionnaire after 3 months of the death.

DETAILED DESCRIPTION:
Patients with advanced cancer report physical, emotional, social and economic problems that may be due to the cancer itself or its treatment. Previous studies have shown the benefit of early palliative care in oncology. However, many Korean patients tend to start palliative care late even in general hospital. Because of the late start of palliative care, the burden of medical expenses increases, on the other hand, the quality of life of terminally ill patients decrease.

In this study, the use of palliative care in advanced cancer patients will be evaluated by a prospective cohort study. The goals of this study are as follow:

First, the clinical, psycho-social, and cognitive factors affecting quality of life, decision making, and hospital utilization (palliative medical team medical treatment, hospice and medical care) of patients with advanced stage cancer will be investigated.

Second, this study will explore the effects of age-specific characteristics on quality of life and care.

Third, an index, which reflects age-specific characteristics and predicts the time and content of terminal care will be developed. Improvements on the quality of life and care of patients with advanced stage of cancer or metastatic cancer are expected to establish effective terminal care strategies through this study.

The patients' symptom and quality of life, choice of medical care, advance care planning and caregiver's burden of care will be evaluated every 3 months after confirming the willingness to use palliative care for cancer patients. 3 months after the death, a caregiver evaluation will be conducted and hospice use, medical expenses will be analyzed.

ELIGIBILITY:
[Adult Patients]

Inclusion Criteria:

* 19 years of age or older and diagnosed as cancer older than 19 years of age
* Stage 4 of advanced Breast Cancer, Colon cancer, gastric cancer, pancreatobiliary cancer, lung cancer, Liver Cancer or Malignant hematologic neoplasm
* Patients under one of the following status : 1) under the standard chemotherapy, 2) interrupted state of standard chemotherapy, 3) under the additional chemotherapy after standard chemotherapy, 4) terminating state of any chemotherapy yet expected to be survive more than 6 months.
* who understand the purpose and method of the study and sign with informed consent form.

Exclusion Criteria:

* who are unable to participate due to poor cognitive capacity
* who cannot read or understand Korean language
* who are unable to complete surveys due to physical conditions

[Pediatric Patients]

Inclusion Criteria:

* Who was diagnosed as pediatric cancer between 0-18 years of age.
* Younger than 30 years of age
* Patients under one of the following status : 1)recurrence after 2nd standard chemotherapy or without remission in leukemia, 2) recurrence after stem cell transplantation, 3) diagnosed as the cancer of poor prognosis : ATRT, glioblastoma multiforme, brainstem glioma etc.
* Patients or their proxy understand the purpose and method of the study and sign with informed consent form.

Exclusion Criteria:

* Parents of patient are unable to participate due to poor cognitive capacity
* Parents of patient do not have legal responsibility or rights of the patient
* Parents of patients cannot speak, read or understand Korean language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced stage of cancer (19 years older) and their families at 14 hospitals nationwide in South Korea
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2016-12-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Overall QOL of EORTC QLQ - Core 15 at 6 months items | Baseline, 3 months, 6 months
  to measure quality of life of adult patients developed by European Organisation for Research and Treatment of Cancer for Palliative Care

SECONDARY OUTCOMES:
Patients survival and Physicians Orders for Life Sustaining Treatment (POLST) documentation | Baseline, 3 months, 6 months
  Patients survival and POLST(Physician Order for Life-Sustaining Treatment) documentation whether patients survive during the study period and write POLST documentation (Since POLST has no legal form in Korea, it is based on the format of each institution.)
Patient Health Questionnaire-9 | Baseline, 3 months, 6 months
  "Patient Health Questionnaire-9 items" is used as assessment tool to measure depression of both patients and their caregivers by completing the questionnaire.
Decision Conflict Scale | Baseline, 6 months
  "Decision Conflict Scale" is used as assessment tool to measure a level of decision conflict in treatment of both patients and their caregivers by completing the questionnaire.
Understanding the illness | Baseline, 3 months, 6 months
  to measure the awareness of patients' status of prognosis in both patients and caregivers through two questions in the questionnaire. The first question is about the idea of the possibility of curing the patient's disease and asks patients thought about whether treatment is available for cure and prolong survival. The second question concerns the life expectancy of the patient.
Self-reported Health Status | Baseline, 3 months, 6 months
  to measure the perceived holistic health status(physical, mental, social, spiritual and general) in both patients and caregivers. caregivers (The patient is asked to answer the perceived health status into five stages.)
KG-7(The Korean Cancer Study Group Geriatric Score) | Baseline, 3 months, 6 months
  To measure Daily functional skills in elderly only in 65-year or order patients.
Medical cost in KRW/person/month | 3 months, 6 months
  Direct medical cost will be collected through National Health Insurance Corporation and Indirect cost will be collected by caregiver's questionnaire. In addition, "EuroQoL 5 Dimensions 5 Levels (EQ-5D-5L)" tool will be included in the patient's questionnaire to measure the condition of patients at the same time.
Utilization of healthcare services | 3 months, 6 months
  In order to analyze the cost effectiveness, investigate the frequency of use of early palliative care programs, the use of life-sustaining treatment and hospicee, and the use of complementary and alternative medicine(CAM). CAM include Chinese medicine, aromatherapy, diet, and yoga, etc.
Preference of Advance care and Palliative care | 3 months, 6 months
  to assess the patient's awareness of advanced care planning and willingness to construct advanced care planning. The preference for palliative care is divided according to the life expectancy. Investigate the preference of palliative care in each case - if the life expectancy is within a year, within a few months, or within a few weeks.
Mcgill Quality of Life (MQOL) | Baseline, 3 months, 6 months
  To measure mental, social, spiritual quality of life of both patients and caregivers
Pediatric Quality of Life Inventory | Baseline, 3 months, 6 months
  "Pediatric Quality of Life Inventory(Peds QL)" will be used as assessment tool for QOL among pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, MD-PhD, Principal Investigator — Seoul National University Hospital
Locations (15):
- South Korea (15):
  - National Cancer Center, Korea, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Daegu Fatima Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Kyunghee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yun JY, Jung JY, Keam B, Lee NR, Kang JH, Kim YJ, Shim HJ, Jung KH, Koh SJ, Ryu H, Yoo SH, Kang E, Yun YH. Depression, performance status, and discontinued treatment mediate an association of curability belief with prognosis in advanced cancer patients. Sci Rep. 2024 Nov 24;14(1):29098. doi: 10.1038/s41598-024-80687-6. PMID 39582048